CLINICAL TRIAL: NCT03974867
Title: Vestibular Prognosis Assessment of the Idiopathic Sudden Sensorineural Hearing Loss With Vestibular Dysfunction Treated With Oral or Intratympanic Glucocorticoids
Brief Title: Vestibular Prognosis Assessment of ISSNHL With Vestibular Dysfunction Treated With Oral or Intratympanic Glucocorticoids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISSNHL RCT
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-06

CONDITIONS: Vestibular Vertigo; Sudden Hearing Loss
Keywords: idiopathic sudden sensorineural hearing loss; vestibular dysfunction; glucocorticoids
MeSH Terms: conditions — Vertigo; Hearing Loss, Sudden | interventions — Prednisone; Methylprednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Prednisone Group (Experimental): 36 participants in Group 1 will receive oral prednisone 1mg/kg/d (maximum daily dosage is no more than 60mg) for 7 days, followed by a 7-day taper.
  Interventions: Drug: Prednisone 5Mg Tab
- Intratympanic Methylprednisolone Group (Experimental): 36 participants in Group 2 will receive 7 intratympanic 40mg/ml methylprednisolone injections in 14 days, one injection every other day.
  Interventions: Drug: Methylprednisolone 40 mg

INTERVENTIONS:
Drug: Prednisone 5Mg Tab — Glucocorticoids:
  d1-d7: Oral Pred. 1mg/kg/d a (maximum daily dosage is no more than 60mg); d8-d9: Oral Pred. 10mg less than d7; d10-d11: Oral Pred. 10mg less than d9; d12: Oral Pred. 10mg less than d11; d13: Oral Pred. 10mg less than d12; d14: Oral Pred. 10mg less than d13;
  Arms: Oral Prednisone Group
Drug: Methylprednisolone 40 mg — Glucocorticoids:
  7 intratympanic injections of 40mg/ml Met. in 14 days, one injection every other day;
  Arms: Intratympanic Methylprednisolone Group

SUMMARY:
Idiopathic sudden sensorineural hearing loss (ISSNHL) is a complicated hearing impairment with unclear etiology and unsatisfying treatment effects. Vestibular dysfunction like vertigo has been considered as a risk factor of profound hearing loss and poor prognosis in ISSNHL. Glucocorticoids, administered through oral or intratympanic way, is currently a regular and standard treatment for ISSNHL based on hearing outcome. However, little investigations have been conducted on recovery process and treatment effects of glucocorticoids on vestibular dysfunctions of ISSNHL. This study aims to evaluate the recovery pattern and possible process of vestibular system in ISSNHL with vestibular dysfunction, and to compare the efficacy of oral or intratympanic glucocorticoids in these participants.

A randomized, outcome assessor- and statistical analyst-blinded, controlled, clinical trial will be carried out. 72 patients complaining of vestibular dysfunction appearing as vertigo, dizziness, imbalance or lateropulsion with ISSNHL will be recruited and randomized into two arms of oral or intratympanic glucocorticoids therapy in 1:1 allocation. The primary outcomes will be subjective feelings evaluated by duration of vestibular dysfunction symptoms, dizziness-related handicap, visual analogue scale for vertigo, and objective vestibular function tests results assessed by sensory organization test, caloric test, video head impulse test and vestibular evoked myogenic potentials. Assessment will be performed at baseline and at 1, 2, 4, and 8 weeks post-randomization.

DETAILED DESCRIPTION:
This study is designed as an 8-week, single-center, randomized, assessor- and analyst-blinded, controlled trial with two parallel interventional groups in a 1:1 allocation.

Patients will be recruited from outpatient clinics of the Eye and ENT Hospital of Fudan University in Shanghai, qualified with well-trained doctors, staff and required facilities for this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 18 to 70 years old;
2. Diagnosed with unilateral ISSNHL according to the National Institute for Deafness and Communication Disorders (NICDC) criteria30: a decrease in hearing of ≥30 decibels (dB), affecting at least 3 consecutive frequencies occurring within a 72-hour period. Since premorbid audiometry is generally unavailable, premorbid hearing level will be defined as the opposite ear's thresholds in this condition;
3. Reported vertigo/dizziness/imbalance/lateropulsion and abnormal results in at least one of the vestibular function tests (including SOT, caloric test, vHIT, cVEMP, and oVEMP);
4. Onset of audio-vestibular symptoms occurred within 7 days;
5. Be willing to sign the informed consent of the study.

Exclusion Criteria:

1. Definite etiologies are found or highly suspected after clinical evaluations, such as vestibular schwannoma, stroke, trauma or demyelinating disease;
2. Diagnosed with a present or previous hearing or balance disorders which might be confused with ISSNHL (history of Meniere's disease, benign paroxysmal positional vertigo, vestibular neuronitis or vestibular migraine; history of otosclerosis; history of luetic, congenital or genetic hearing loss, etc.);
3. Hearing level (evaluated with PTA) in the unaffected ear is abnormal, so that a premorbid hearing level of the affected ear may not be estimated;
4. Suspected as central vestibular dysfunction, evaluated by present and previous medical history, physical examination and VNG;
5. Present with conditions contraindicated systemic glucocorticoids use, such as tuberculosis, hepatitis C or B infection, active herpes zoster infection or other known human immunodeficiency virus, pancreatitis, insulin-dependent diabetes mellitus, severe osteoporosis, chronic renal insufficiency or gastrointestinal ulcer;
6. A history of more than 3 days sufficient systemic glucocorticoids uses (≥1 mg/kg/d) within 3 months which may increase the risk of adverse effects. Considering that the glucocorticoids is a well-acknowledged standard treatment and that the patients might have probably received initial systemic glucocorticoids in emergency before outpatient appointment, we only excluded those who have received sufficient glucocorticoids (≥1mg/kg/d prednisone) for more than 3 days in previous 3 months;
7. Having received other systemic etiological treatments for ISSNHL (including hyperbaric oxcygen therapy (HBOT), thrombolytic drugs and antiviral drugs) which may confound the effects of study drugs. Patients who received only emergency or symptomatic treatments will not be excluded (i.e., betahistine, promethazine, diazepam, mecobalamin or ginkgo biloba leaves extracts);
8. Not appropriate for receiving vestibular function tests due to combination of fracture, inflammatory or suppurative ear disease, severe cervical spondylosis or severe psychotic disorders;
9. Multiple organ dysfunction or unstable vital signs;
10. Pregnancy or lactation;
11. Evaluated as unsuitable for the trial for any other reasons by investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Complete recovery rates of vestibular function tests within 8 weeks | 8 weeks from baseline
  To evaluate the recovery of vestibular function and subjective vestibular dysfunction feelings, we set the recovery rates of the whole battery of vestibular function tests (SOT/caloric test/vHIT/VEMPs) as the primary outcome, which is the proportion of patients whose abnormal results of vestibular function tests at baseline recover to normal during the 8-weeks follow-up:
  recovery rate (8 weeks)=(number of patients recover from abnormal result at baseline to normal during at 8-weeks follow-up)/(number of all enrolment participants patients with abnormal result at baseline)×100%;

SECONDARY OUTCOMES:
Change of SOT vestibular scores at 4-week follow-up | 4 weeks from baseline
  Change of the vestibular scores in SOT at 4-week follow-up from baseline
Change of SOT vestibular scores at 8-week follow-up | 8 weeks from baseline
  Change of the vestibular scores in SOT at 8-week follow-up from baseline
Change of unilateral weakness of caloric test at 4-week follow-up | 4 weeks from baseline
  Change of unilateral weakness (UW) of caloric test at 4-week follow-up
Change of unilateral weakness of caloric test at 8-week follow-up | 8 weeks from baseline
  Change of UW of caloric test at 8-week follow-up
Recovery rate of vHIT at 4-week follow-up | 4 weeks from baseline
  Recovery rate of vHIT at 4-week follow-up
Recovery rate of vHIT at 8-week follow-up | 8 weeks from baseline
  Recovery rate of vHIT at 8-week follow-up
Recovery rate of cVEMP at 4-week follow-up | 4 weeks from baseline
  Recovery rate of cVEMP at 4-week follow-up
Recovery rate of cVEMP at 8-week follow-up | 8 weeks from baseline
  Recovery rate of cVEMP at 8-week follow-up
Recovery rate of oVEMP at 4-week follow-up | 4 weeks from baseline
  Recovery rate of oVEMP at 4-week follow-up
Recovery rate of oVEMP at 8-week follow-up | 8 weeks from baseline
  Recovery rate of oVEMP at 8-week follow-up
Change of PTA at 1 week from baseline | 1 week
  change of average of PTA from baseline at 1-week follow-up
Change of PTA at 2 week from baseline | 2 weeks
  change of average of PTA from baseline at 2-weeks follow-up
Change of PTA at 4 week from baseline | 4 weeks
  change of average of PTA from baseline at 4-weeks follow-up
Change of PTA at 8 week from baseline | 8 weeks
  change of average of PTA from baseline at 8-weeks follow-up
Change of score of VAS for tinnitus (VAS-T) at 1 week from baseline | 1 weeks
  Change of scores of VAS-T from baseline at 1-week follow-up. Visual Analogue Scale for Tinnitus (VAS-T) is a universal psychometric scale evaluating subjective tinnitus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.
Change of score of VAS for vertigo (VAS-V) at 1 week from baseline | 1 weeks
  Change of scores of VAS-V from baseline at 1-week follow-up. Visual Analogue Scale for Tinnitus (VAS-T) is a universal psychometric scale evaluating subjective tinnitus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.
Change of score of VAS-T at 2 week from baseline | 2 weeks
  Change of scores of VAS-T from baseline at 2-weeks follow-up. Visual Analogue Scale for Tinnitus (VAS-T) is a universal psychometric scale evaluating subjective tinnitus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.
Change of score of VAS-V at 2 week from baseline | 2 weeks
  Change of scores of VAS-V from baseline at 2-weeks follow-up. Visual Analogue Scale for Tinnitus (VAS-T) is a universal psychometric scale evaluating subjective tinnitus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.
Change of score of VAS-T at 4 week from baseline | 4 weeks
  Change of scores of VAS-T from baseline at 4-weeks follow-up. Visual Analogue Scale for Tinnitus (VAS-T) is a universal psychometric scale evaluating subjective tinnitus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.
Change of score of VAS-V at 4 week from baseline | 4 weeks
  Change of scores of VAS-V from baseline at 4-weeks follow-up. Visual Analogue Scale for Tinnitus (VAS-T) is a universal psychometric scale evaluating subjective tinnitus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.
Change of score of VAS-T at 8 week from baseline | 8 weeks
  Change of scores of VAS-T from baseline at 8-weeks follow-up. Visual Analogue Scale for Tinntius (VAS-T) is a universal psychometric scale evaluating subjective tinnitus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.
Change of score of VAS-V at 8 week from baseline | 8 weeks
  Change of scores of VAS-V from baseline at 8-weeks follow-up. Visual Analogue Scale for Tinntius (VAS-T) is a universal psychometric scale evaluating subjective tinnitus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Huawei Li, MD, PhD, Study Chair — Eye and ENT Hospital of Fudan University
Locations (1):
- Otorhinolaryngology Department, Eye and ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stachler RJ, Chandrasekhar SS, Archer SM, Rosenfeld RM, Schwartz SR, Barrs DM, Brown SR, Fife TD, Ford P, Ganiats TG, Hollingsworth DB, Lewandowski CA, Montano JJ, Saunders JE, Tucci DL, Valente M, Warren BE, Yaremchuk KL, Robertson PJ; American Academy of Otolaryngology-Head and Neck Surgery. Clinical practice guideline: sudden hearing loss. Otolaryngol Head Neck Surg. 2012 Mar;146(3 Suppl):S1-35. doi: 10.1177/0194599812436449. PMID 22383545
- [Background] Rauch SD, Halpin CF, Antonelli PJ, Babu S, Carey JP, Gantz BJ, Goebel JA, Hammerschlag PE, Harris JP, Isaacson B, Lee D, Linstrom CJ, Parnes LS, Shi H, Slattery WH, Telian SA, Vrabec JT, Reda DJ. Oral vs intratympanic corticosteroid therapy for idiopathic sudden sensorineural hearing loss: a randomized trial. JAMA. 2011 May 25;305(20):2071-9. doi: 10.1001/jama.2011.679. PMID 21610239
- [Background] Yu H, Li H. Association of Vertigo With Hearing Outcomes in Patients With Sudden Sensorineural Hearing Loss: A Systematic Review and Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2018 Aug 1;144(8):677-683. doi: 10.1001/jamaoto.2018.0648. PMID 29931169
- [Background] Yu H, Li H. Vestibular Dysfunctions in Sudden Sensorineural Hearing Loss: A Systematic Review and Meta-analysis. Front Neurol. 2018 Feb 5;9:45. doi: 10.3389/fneur.2018.00045. eCollection 2018. PMID 29459846
- [Derived] Hao W, Zhao L, Yu H, Li H. Vestibular prognosis in idiopathic sudden sensorineural hearing loss with vestibular dysfunction treated with oral or intratympanic glucocorticoids: a protocol for randomized controlled trial. Trials. 2020 Jul 22;21(1):669. doi: 10.1186/s13063-020-04579-6. PMID 32698830